CLINICAL TRIAL: NCT04183465
Title: Effectiveness of an Early, Tailored, Physical Activity Intervention in ELderly Patients With Myocardial INfarction: the PIpELINe Randomized Clinical Trial
Brief Title: Physical Activity Intervention in ELderly Patients With Myocardial INfarction
Acronym: PIpELINe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Azienda Usl di Bologna (Other Government); Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Full Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 376/2019/Sper/AOUFe
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Aging
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The members of the Clinical Event Committee will be blinded to randomization arm during all phases of the adjudications of the adverse events
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education (Active Comparator): All patients randomized to health education received a single in-person visit, one month post discharge, which included a 30-minute counselling session, supported by educational materials and tailoring of the medical treatment. The educational material provided standardized recommendations on diet, smoking cessation, and physical activity. Quality of life, functional capacity and home physical activity are assessed by proper tools.
  Interventions: Other: Health Education
- Multi-domain lifestyle intervention (Experimental): All patients randomized to experimental arm will receive diet counselling, aggressive control of CV risk factors, smoke cessation program and exercise training. The physical activity (PA) intervention will start the program with a supervised PA session immediately after the inclusion visit. Quality of life, functional capacity and daily activities will be assessed by proper tools. The program provides 6 supervised PA sessions (30, 60, 90, 180, 270 and 360 days after hospital discharge [T0]). At the end of each supervised session, calisthenics exercises derived from Otago Exercise Program are prescribed.
  Interventions: Other: Multi-domain lifestyle intervention

INTERVENTIONS:
Other: Health Education — Current gold standard in older patients admitted to hospital for MI. The group will receive a 20-minute session with one of the study physicians. Both the patient and relatives will attend these sessions. The study physician will stress the major issues related to a heart-healthy lifestyle and will explain the importance of PA as a powerful and independent factor to improve cardiovascular health and minimize cardiovascular risk. A detailed brochure explaining the benefits of physical activity will be provided to all patients
  Arms: Health Education
Other: Multi-domain lifestyle intervention — The intervention includes diet counselling, smoke cessation program, aggressive CV risk control and PA intervention. The PA intervention consisted of supervised sessions combined with an individualized home-based PA program. Centre-based sessions will be supervised by a sports physician and a nurse, and will take approximately 30 to 40 minutes, including a moderate standardized treadmill-walk, and strength and balance exercises. Based on the practice sessions, patients will receive a walking program to perform at home, unsupervised. The PA programs will be individualized, and consistent with current international recommendations. A selection of calisthenic exercises will be prescribed. Participants will be encouraged to perform the exercises three times per week (approximately 20 minutes). Adjustment of the type and intensity of the home-based PA regimen will be made at each visit. The PA program will be extensively described to the patient and family members.
  Arms: Multi-domain lifestyle intervention

SUMMARY:
Elderly patients presenting with myocardial infarction (MI) are the highest risk population with the worst prognosis. No trial has ever been designed to optimize their outcome through a systematic improvement of their physical performance. Cardiac rehabilitation demonstrated to improve prognosis of patients after MI. However, real-life data shows that older patients are not referred to rehabilitation centers or they have low rate of attendance because of the high number of rehabilitation sessions and of logistic problems. So, data about effectiveness of rehabilitation programs in older MI patients is lacking.

The "Physical Activity Intervention for Elderly Patients with Reduced Physical Performance after acute coronary syndrome (HULK)" pilot study (NCT03021044) enrolled older MI patients and it demonstrated the feasibility and effectiveness of an early, tailored and low-cost physical activity intervention in terms of physical performance assessed by Short Physical Performance Battery (SPPB) score, that is strongly related to prognosis. The HULK study was focused on exercise training and not powered for hard endpoints. If a multi-domain lifestyle intervention in an adequately powered study may further improve prognosis is unknown. Thus, the investigator's hypothesis for the PIpELINe trial is that an early, tailored and low-cost multi-domain lifestyle intervention may improve prognosis of older MI patients compared to health education alone. The primary outcome is a composite of 1-year cardiovascular death and hospital readmission for cardiovascular cause.

DETAILED DESCRIPTION:
The PIpELINe trial will include older MI patients. All patients aged 65 years and older undergoing coronary angiography because of MI must be screened for eligibility. Patient's eligibility must be assessed after percutaneous revascularization of all lesions considered susceptible of treatment. After verifying inclusion and exclusion criteria and after eligibility is confirmed, written informed consent must be obtained prior to randomization. At the time of the discharge (T0) SPPB test will be performed; in case of a score between 4 and 9, the patient will be evaluated 1-month after discharge at the inclusion visit (T1). If SPPB value is confirmed to be between 4 and 9, randomization will be performed. Key baseline patient characteristics (i.e., inclusion/exclusion criteria, demographics, medical history, details of cardiovascular anatomy and of revascularization, ECG and laboratory test results, echocardiographic data during the index hospitalization) will be recorded on the electronic Case Report Forms (eCRF). All angiographic and echocardiographic data will be collected and forwarded to a core lab for further assessment.

Randomization will be performed during the inclusion visit (T1), 30 days after discharge. Randomization will be performed centrally using an internet-based system. The patient identification number (Patient ID) and the treatment allocation will be assigned by the central randomization system. Patients will be randomized to physical activity group or health education group by a 2:1 allocation. Treatment allocation will be assigned according to a computer-generated randomization list stratified by center. All randomized patients are irrevocably in the study, whether or not they are subsequently found to be eligible, or actually receiving the allocated treatment. Therefore, all patients must be followed until the pre-specified study end date.

The aim of the study is to demonstrate that the proposed multi-domain lifestyle intervention reduces the composite endpoint of cardiovascular death and hospital readmission for cardiovascular cause. The primary endpoint is at 1 year. The follow-up will be extended up to 2 and 3 years.

The protocol includes 3 pre-specified substudies. The possibility to participate in the substudy is left to patient's decision and doesn't preclude the procedures of the main protocol.

* Anxiety and depression: previous studies reported an association between cardiovascular events and a subsequent appearance of mood disorders which could determine a lack in following secondary prevention recommendations. No data is available about these disorders in older adults. In order to assess depression after MI in older patients and the effect of physical activity intervention on mood disorders, this sub-study will be performed.
* Mitochondrial function: in both study groups the mitochondrial functional are investigated starting from blood samples and skin biopsy. Skin biopsy is performed to obtain fibroblasts. In-vitro assessment of the mitochondrial function is done on the fibroblasts of patients. The parameters obtained are related with the effectiveness of physical intervention and with the benefit obtained. A total of at least 30 patients is required.
* Lymphocyte and miRNA activity: taking into account the immunosenescence and the benefits of physical activity on the immune system, this sub-study aims to obtain data regarding T-lymphocyte function in older adults and to assess the effect of physical activity intervention on the function of the different groups of T-lymphocyte. Analyses of physical activity effects on micro ribonucleic acids (miRNAs) are also performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥65 years
* Hospital admission for myocardial infarction
* Invasive management during index hospitalization including coronary artery angiography (± percutaneous coronary revascularization)
* SPPB value 4-9 at 1-month visit after hospital discharge
* Informed consent

Exclusion Criteria:

1. Multivessel coronary artery disease or left main coronary artery disease candidate to surgical revascularization
2. Planned staged percutaneous coronary intervention (PCI)
3. Non-cardiovascular co-morbidity reducing life expectancy to < 1 year
4. Any factor precluding 1-year follow-up
5. Severe aortic or mitral disease
6. Ejection fraction <30%
7. Chronic heart failure New York Heart Association (NYHA) III-IV
8. Severe cognitive impairment (SPMSQ <4)
9. Impossibility to do physical activity due to physical impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 512 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative occurrence of cardiovascular death and hospital readmission for cardiovascular cause | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of 1-year composite endpoint of cardiovascular death plus hospital readmission for cardiovascular cause.

SECONDARY OUTCOMES:
Cumulative occurrence of all-cause death | 1-year
  To test the superiority of the early and tailored physical activity intervention over the health education alone in terms of all-cause death
Cumulative occurrence of all-cause death | 3-year
  To test the superiority of the early and tailored physical activity intervention over the health education alone in terms of all-cause death
Cumulative occurrence of cardiovascular death | 1-year
  To test the superiority of the early and tailored physical activity intervention over the health education alone in terms of cardiovascular death
Cumulative occurrence of cardiovascular death | 3-year
  To test the superiority of the early and tailored physical activity intervention over the health education alone in terms of cardiovascular death
Cumulative occurrence of hospital readmission for cardiovascular cause | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for cardiovascular cause.
Cumulative occurrence of hospital readmission for cardiovascular cause | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of composite endpoint of hospital readmission for cardiovascular cause.
Cumulative occurrence of cardiovascular death and hospital readmission for cardiovascular cause | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of composite endpoint of cardiovascular death plus hospital readmission for cardiovascular cause.
Cumulative occurrence of hospital readmission for heart failure | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for heart failure
Cumulative occurrence of hospital readmission for heart failure | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for heart failure
Cumulative occurrence of hospital readmission for myocardial infarction | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for myocardial infarction
Cumulative occurrence of hospital readmission for myocardial infarction | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for myocardial infarction
Cumulative occurrence of hospital readmission for coronary revascularization | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for coronary revascularization
Cumulative occurrence of hospital readmission for coronary revascularization | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for coronary revascularization
Cumulative occurrence of cerebrovascular accident | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of cerebrovascular accident
Cumulative occurrence of cerebrovascular accident | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of cerebrovascular accident
Cumulative occurrence of hospital readmission for any cause | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for any cause
Cumulative occurrence of hospital readmission for any cause | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for any cause
Cumulative occurrence of hospital readmission for any non-cardiovascular cause | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for any non-cardiovascular cause
Cumulative occurrence of hospital readmission for any non-cardiovascular cause | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of hospital readmission for any non-cardiovascular cause
Cumulative occurrence of bleeding adverse events | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of bleeding adverse events
Cumulative occurrence of bleeding adverse events | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of bleeding adverse events

OTHER OUTCOMES:
Short Physical Performance Battery | 6-month
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (SPPB ranges from 0 to 12, higher values mean better physical performance)
Short Physical Performance Battery | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (SPPB ranges from 0 to 12, higher values mean better physical performance)
Short Physical Performance Battery | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (SPPB ranges from 0 to 12, higher values mean better physical performance)
Handgrip strength | 6-month
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (handgrip strength, ranges from 0 to infinity, higher values mean better physical performance)
Handgrip strength | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (handgrip strength, ranges from 0 to infinity, higher values mean better physical performance)
Handgrip strength | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (handgrip strength, ranges from 0 to infinity, higher values mean better physical performance)
Gait speed | 6-month
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (10 meters gait speed ranges from 0 to infinity, higher values mean better physical performance)
Gait speed | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (10 meters gait speed ranges from 0 to infinity, higher values mean better physical performance)
Gait speed | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of physical performance (10 meters gait speed ranges from 0 to infinity, higher values mean better physical performance)
EQ5D visual analogue scale | 6-month
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of quality of life (EQ5D VAS points)
EQ5D visual analogue scale | 1-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of quality of life (EQ5D VAS points)
EQ5D visual analogue scale | 3-year
  To assess the superiority of the early and tailored physical activity intervention over health education alone in terms of quality of life (EQ5D VAS points)

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Medicina dello Sport SSD, Bologna, BO
  - Centro Studi Biomedici applicati allo Sport, Ferrara, Ferrara, FE
  - Ospedale Guglielmo da Saliceto, Piacenza, Piacenza, PC
  - UO Cardiologia, Ospedale Maggiore, Bologna
  - Cardiology Unit, Ferrara
  - Cardiologia Riabilitativa, AUSL d Ferrara, Lagosanto
  - Medicina dello Sport, AUSL Piacenza, Piacenza

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: After publication of the main findings
Access Criteria: It will be necessary a formal request to the Executive Committee of the study. The request will be analyzed and considered for acceptance

REFERENCES:
- [Result] Tonet E, Raisi A, Zagnoni S, Chiaranda G, Pavasini R, Vitali F, Gibiino F, Campana R, Boccadoro A, Scala A, Canovi L, Amantea V, Matese C, Berloni ML, Piva T, Zerbini V, Cardelli LS, Pasanisi G, Mazzoni G, Casella G, Grazzi G, Campo G. Multi-domain lifestyle intervention in older adults after myocardial infarction: rationale and design of the PIpELINe randomized clinical trial. Aging Clin Exp Res. 2023 May;35(5):1107-1115. doi: 10.1007/s40520-023-02389-9. Epub 2023 Mar 25. PMID 36964866
- [Derived] Tonet E, Raisi A, Zagnoni S, Chiaranda G, Pasanisi G, Aschieri D, D'Intino PE, Pavasini R, Cimaglia P, Campana R, Vitali F, Piva T, Casella G, Caglioni S, Zerbini V, Bugani G, Cocco M, Menegatti E, De Raffele M, Mandini S, Martella D, Pesenti N, Mazzoni G, Biscaglia S, Volpato S, Grazzi G, Campo G; PIpELINe Trial Investigators. Multidomain Rehabilitation for Older Patients with Myocardial Infarction. N Engl J Med. 2025 Sep 11;393(10):973-982. doi: 10.1056/NEJMoa2502799. Epub 2025 Aug 29. PMID 40879431